CLINICAL TRIAL: NCT01503515
Title: A Phase III Open-Label Trial of Caspofungin vs. Azole Prophylaxis for Patients at High-Risk for Invasive Fungal Infections (IFI) Following Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Caspofungin Acetate, Fluconazole, or Voriconazole in Preventing Fungal Infections in Patients Following Donor Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACCL1131; NCI-2012-00102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000721415; ACCL1131 (Other: Children's Oncology Group); COG-ACCL1131 (Other: DCP); ACCL1131 (Other: CTEP); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Fungal Infection; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Mycoses; Hematologic Neoplasms | interventions — Caspofungin; Fluconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Arm I (caspofungin acetate) (Experimental): Patients receive caspofungin acetate IV over 1 hour once daily (QD) beginning within 24 hours of allogeneic HSCT (day -1 or 0) and continuing until day 42 in the absence of invasive fungal infections or disease progression.
  Interventions: Drug: Caspofungin Acetate; Other: Laboratory Biomarker Analysis
- Arm II (fluconazole or voriconazole) (Active Comparator): Patients receive fluconazole IV over 1-2 hours QD or PO QD; or voriconazole IV over 1-2 hours QD or PO BID beginning within 24 hours of allogeneic HSCT (day -1 or 0) and continuing until day 42 in the absence of invasive fungal infections or disease progression.
  Interventions: Drug: Fluconazole; Other: Laboratory Biomarker Analysis; Drug: Voriconazole

INTERVENTIONS:
Drug: Caspofungin Acetate — Given IV
  Other Names: Cancidas
  Arms: Arm I (caspofungin acetate)
Drug: Fluconazole — Given IV or PO
  Other Names: Diflucan
  Arms: Arm II (fluconazole or voriconazole)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Voriconazole — Given IV or PO
  Other Names: Vfend
  Arms: Arm II (fluconazole or voriconazole)

SUMMARY:
This randomized phase III trial studies how well caspofungin acetate works compared to fluconazole or voriconazole in preventing fungal infections in patients following donor stem cell transplant. Caspofungin acetate, fluconazole, and voriconazole may be effective in preventing fungal infections in patients following donor stem cell transplant. It is not yet known whether caspofungin acetate is more effective than fluconazole or voriconazole in preventing fungal infections in patients following donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if caspofungin (caspofungin acetate) is associated with a lower incidence of proven/probable invasive fungal infections (IFI) during the first 42 days following allogeneic hematopoietic cell transplantation (HCT) at high-risk for IFI compared with azole (fluconazole or voriconazole) prophylaxis.

EXPLORATORY OBJECTIVES:

I. To determine if caspofungin is associated with a lower incidence of proven/probable IFI during the first 100 days following high-risk allogeneic HCT compared with azole (fluconazole or voriconazole) prophylaxis. (Exploratory) II. To determine if caspofungin is associated with a lower incidence of proven/probable IFI during the first 42 and 100 days following high-risk allogeneic HCT compared with fluconazole prophylaxis. (Exploratory) III. To determine if caspofungin is associated with a lower incidence of proven/probable IFI during the first 42 and 100 days following high-risk allogeneic HCT compared with voriconazole prophylaxis. (Exploratory) IV. To determine if caspofungin is associated with a superior fungal-free survival (FFS) (time to death or proven/probable IFI) at 42 and 100 days following high-risk allogeneic HCT compared with azole prophylaxis. (Exploratory) V. To describe the effect that caspofungin and azoles have on the incidence and severity of acute graft-versus-host disease (GVHD). (Exploratory) VI. To define the test characteristics of weekly Fungitell assay testing for identifying IFI in pediatric hematopoietic stem cell transplantation (HSCT) recipients receiving antifungal prophylaxis during the post-transplant neutropenic period. (Exploratory) VII. To create a deoxyribonucleic acid (DNA) specimen bank in anticipation of the development of biology correlative studies exploring the relationship between IFI and single nucleotide polymorphisms (SNPs) of genes involved in immunity. (Exploratory)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive caspofungin acetate intravenously (IV) over 1 hour once daily (QD) beginning within 24 hours of allogeneic HSCT (day -1 or 0) and continuing until day 42 in the absence of invasive fungal infections or disease progression.

ARM II: Patients receive fluconazole IV over 1-2 hours QD or orally (PO) QD; or voriconazole IV over 1-2 hours QD or PO twice daily (BID) beginning within 24 hours of allogeneic HSCT (day -1 or 0) and continuing until day 42 in the absence of invasive fungal infections or disease progression.

After completion of study treatment, patients are followed up until day 100.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * For centers that will use fluconazole as the antifungal comparator:

    * Age >= 3 months and < 21 years
  * For centers that will use voriconazole as the antifungal comparator:

    * Age >= 2 years and < 21 years
* The patient must be undergoing allogeneic HCT from any donor (including matched related) with any stem cell source for any underlying condition
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin < 2.5 mg/dL unless the increase in bilirubin is attributable to Gilbert's syndrome
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 5 x upper limit of normal (ULN) for age
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Within 90 days of enrollment:

  * Patients with a proven or probable invasive mold infection are not eligible
  * Patients with an incompletely treated invasive yeast infection are not eligible
  * Patients with an elevated galactomannan level (>= 0.5 index) within 30 days prior to time of enrollment (if performed) must have a full evaluation for invasive aspergillosis (including a negative chest computed tomography [CT] scan) during that time period to be eligible for enrollment
* Patients receiving treatment for an IFI are not eligible
* Patients with a history of echinocandin or azole hypersensitivity are not eligible
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation
* Lactating females are not eligible unless they have agreed not to breastfeed their infants

Ages: 3 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 292 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Dvorak, Principal Investigator — Children's Oncology Group
Locations (49):
- United States (46):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Dvorak CC, Fisher BT, Esbenshade AJ, Nieder ML, Alexander S, Steinbach WJ, Dang H, Villaluna D, Chen L, Skeens M, Zaoutis TE, Sung L. A Randomized Trial of Caspofungin vs Triazoles Prophylaxis for Invasive Fungal Disease in Pediatric Allogeneic Hematopoietic Cell Transplant. J Pediatric Infect Dis Soc. 2021 Apr 30;10(4):417-425. doi: 10.1093/jpids/piaa119. PMID 33136159
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole or Voriconazole)
Started | 145 | 147
Completed | 124 | 112
Not Completed | 21 | 35
Not completed — Adverse Event | 4 | 5
Not completed — Death | 0 | 1
Not completed — Physician Decision | 14 | 23
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Institutional dx of proven/probable IFI | 2 | 4
Not completed — Ineligible | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole or Voriconazole) | Total
Number analyzed (Participants) | 145 | 147 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 134 | 133 | 267
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (5.7) | 9.1 (6.0) | 9.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 89 | 91 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 113 | 107 | 220
  Unknown or Not Reported | 6 | 13 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 9 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 22 | 33
  White | 110 | 97 | 207
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 11 | 20 | 31
Region of Enrollment [Number; unit: participants]
  United States | 136 | 132 | 268
  Canada | 9 | 15 | 24

OUTCOME MEASURES:

1. Primary Outcome: 42-day-cumulative Incidence of Proven or Probable Invasive Fungal Infections (IFI)
Description: Kaplan-Meier curves will be used to estimate the 42- day-cumulative incidence of proven/probable IFI following allogeneic HCT for patients randomized to the 2 arms. Proven or probable IFI is defined according to criteria developed by the European Organization for Research and Treatment of Cancer (EORTC)/Mycoses Study Group (MSG).
Time Frame: Up to 42 days following allogeneic HCT
Population: study enrolled 292 patients (145 randomized to caspofungin and 147 randomized to an azole) . Two patients (1 caspofungin, 1 azole) were ineligible, resulting in 290 patients (144 caspofungin, 146 azole) included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole or Voriconazole)
Number analyzed (Participants) | 144 | 146
percentage of patients | 1.4 [0.3 to 5.4] | 1.4 [0.4 to 5.5]

2. Other Pre Specified Outcome: 100-day-cumulative Incidence of Proven or Probable IFI
Description: Kaplan-Meier curves will be used to estimate the 100- day-cumulative incidence of proven/probable IFI following allogeneic HCT for patients randomized to the 2 arms. Proven or probable IFI is defined according to criteria developed by the European Organization for Research and Treatment of Cancer (EORTC)/Mycoses Study Group (MSG).
Time Frame: Up to day 100 following allogeneic HCT
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Fungal-free-survival
Description: Defined as time to death or proven/probable IFI during the first 42 days following allogeneic HCT.
Time Frame: Up to 42 days following allogeneic HCT
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Incidence of Overall Clinical GVHD Grades III and IV
Description: The percentage distribution of overall clinical grades III and IV will be estimated for each arm.
Time Frame: Up to 100 days after allogeneic HCT
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Incidence of Overall Clinical GVHD Grades II to IV
Description: The percentage distribution of overall clinical grades II and IV will be estimated for each arm.
Time Frame: Up to 100 days after allogeneic HCT
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Fungal-free-survival
Description: Defined as time to death or proven/probable IFI during the first 100 days following allogeneic HCT.
Time Frame: Up to 100 days following allogeneic HCT
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Sensitivity of Beta-D Glucan Assay for the Diagnosis of IFI Using Fungitell Assay
Description: Sensitivity of the beta-D glucan assay will be determined using standard formulas and EORTC/MSG criteria as the gold standard.
Time Frame: Up to day 42 following allogeneic HCT
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Specificity of Beta-D Glucan Assay for the Diagnosis of IFI Using Fungitell Assay
Description: Specificity of the beta-D glucan assay will be determined using standard formulas and EORTC/MSG criteria as the gold standard.
Time Frame: Up to day 42 following allogeneic HCT
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Positive Predictive Value of Beta-D Glucan Assay for the Diagnosis of IFI Using Fungitell Assay
Description: Positive predictive value of the beta-D glucan assay will be determined using standard formulas and EORTC/MSG criteria as the gold standard.
Time Frame: Up to day 42 following allogeneic HCT
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Negative Predictive Value of Beta-D Glucan Assay for the Diagnosis of IFI Using Fungitell Assay
Description: Negative predictive value of the beta-D glucan assay will be determined using standard formulas and EORTC/MSG criteria as the gold standard.
Time Frame: Up to day 42 following allogeneic HCT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Collected Adverse Events within the 100 day observation period
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole or Voriconazole)
All-Cause Mortality (participants affected / at risk) | 9/144 | 10/146
Serious Adverse Events (participants affected / at risk) | 4/144 | 3/146
Other Adverse Events (participants affected / at risk) | 29/144 | 30/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Caspofungin Acetate) (N=144) | Arm II (Fluconazole or Voriconazole) (N=146)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Caspofungin Acetate) (N=144) | Arm II (Fluconazole or Voriconazole) (N=146)
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 5
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
GGT increased (Investigations) | 4 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 1
Multi-organ failure (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT01503515/Prot_SAP_ICF_000.pdf